CLINICAL TRIAL: NCT00787436
Title: Secondary Prophylaxis of Gastrointestinal Bleeding in Cirrhotic Patients Using Thalidomide
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CEL-20237; IRB00000536; FWA00005367; 34-0714585; OSR-20070905-01
Record Dates: First submitted 2008-11-05; First posted 2008-11-07 (Estimated); Last update posted 2013-07-31 (Estimated); Status verified 2013-07

CONDITIONS: Gastrointestinal Hemorrhage; Portal Hypertension
Keywords: portal hypertension; Gastroesophageal; Varices; Liver disease; cirrhosis
MeSH Terms: conditions — Gastrointestinal Hemorrhage; Hypertension, Portal; Varicose Veins; Liver Diseases; Fibrosis | interventions — Thalidomide; Propranolol; Nadolol; Timolol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (No Intervention): Standard of care with normal treatment
- Thalidomide (Active Comparator): Standard of care and treatment using Thalidomide
  Interventions: Drug: Thalidomide

INTERVENTIONS:
Drug: Thalidomide — Medical therapy has been used to decrease upper gastrointestinal bleeding in cirrhotics Non Selective beta blockers have been shown to effectively decrease the portal venous pressure
  Other Names: propranolol; nadolol; timolol
  Arms: Thalidomide

SUMMARY:
The natural history of cirrhosis has a symptomatic and asymptomatic stage. The symptoms include the development of ascites, hepatic encephalopathy, or variceal bleeding. The development of portal hypertension represents a critical transition point in the natural history of cirrhosis, contributing to, or directly responsible for all of these events. It is defined by an increase in intrahepatic vascular resistance to portal venous inflow, with the subsequent development of collateral vessels, such as esophageal or gastric varices. As portal pressures rise over time, however, the resulting increase in variceal size and wall tension translates into an increasing likelihood of rupture and bleeding, leading to death in about 30% of patients. Over the last twenty years, data have emerged regarding the role of tumor necrosis factor (TNFα) in portal hypertension from animal models as well as in vitro experiments. Portal hypertension is a condition characterized by vasodilatation and a hyperdynamic circulation, driven by relative overproduction of nitric oxide23. In animal trials using inhibitors of TNF it has been shown to decrease the development of the hyperdynamic circulatory state and portal pressure.24-25 Based on these data, investigators have examined the role of TNF inhibition with thalidomide. Significant improvement in blocking the development of the hyperdynamic circulation and portal pressures was demonstrated.26 Human trials have also show the efficacy of thalidomide in reducing portal pressures. In that these trials have shown promising results further investigation is

DETAILED DESCRIPTION:
Treatment duration with thalidomide will be for 16 weeks, beginning in the hospital setting immediately after the index bleed, and clinical follow-up additional six months. Follow-up in both the hepatology, outpatient clinic area and the endoscopy suite will occur. Step wise thalidomide dosing will be 100 mg/d once a day at night. If no evidence of toxicity is noted after 5 doses, the dose will be increased to 200 mg/d, and continued on that dose as an outpatient until completion of the study protocol at 16 weeks. Patients will be followed daily while inpatients, and subsequently at two-week intervals upon discharge. Females of child-bearing potential will be seen weekly for the first month and must have a confirmed negative pregnancy test prior to being dispensed the next one week supply of study drug. After the first month, females of child-bearing potential will be seen every two weeks as will all other subjects. Standard follow-up medical care after esophageal variceal bleeding in patients who have undergone endoscopic therapy will include:

follow-up endoscopy at regular intervals until variceal obliteration, using either endoscopic variceal ligation (EVL) or sclerotherapy titrated dose of a nonselective beta blocker (propranolol).

At each follow-up visit, patients will be assessed for development of any interim outcome of interest:

overt upper gastrointestinal bleeding need for transfusion worsening clinical status

Patients will initially be followed daily while hospitalized. outpatient visits will occur every two-week intervals upon discharge. Standard follow-up medical care after esophageal variceal bleeding in patients who have undergone endoscopic therapy will include:

follow-up endoscopy at regular intervals until variceal obliteration, using either endoscopic variceal ligation (EVL) or sclerotherapy titrated dose of a nonselective beta blocker (propranolol).

At each follow-up visit, patients will be assessed for development of any interim outcome of interest:

overt upper gastrointestinal bleeding need for transfusion worsening clinical status the need for TIPS, liver transplantation or death. In addition, patients and their families will be questioned for any evidence of potential toxicity as assessed by using the CTC Toxicity grade version 3, or adverse outcomes by one of the study investigators as well as a nurse coordinator, using a standardized questionnaire along with a regular clinical

ELIGIBILITY:
Inclusion Criteria:

* Endoscopic confirmation or portal hypertension related GI bleeding
* Over the age of 18 with the ability to willingly sign an informed consent
* Adequate performance status and cognitive ability
* Patients must be willing to comply with all FDA-mandated prescribing and safety while taking Thalidomide
* Hemodynamically stable with no evidence of ongoing bleeding (defined as a Hgb that has not varied by more than 10% over 12 hour period.)

Exclusion Criteria:

* No other serious illness or medical condition including unstable cardiac disease requiring treatment, new onset crescendo or rest angina. Stable exertional angina is acceptable.
* No history of significant neurological or psychiatric disorders including psychotic disorders, dementia, or seizures or active infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2006-05; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
The proposed study would use a novel approach to prophylaxis, using thalidomide, an oral TNF inhibitor, in conjunction with a betablocker to prevent rebleeding of upper gastrointestinal bleeding in patients with cirrhosis and portal hyperte | 16 week duration

SECONDARY OUTCOMES:
The secondary endpoint is to examine the impact on progression of liver disease in this population, including development of other complications of chronic liver disease, such as encephalopathy, hepatorenal syndrome and patient survival | 16 week duration

CONTACTS AND LOCATIONS:
Locations (1):
- Cleveland Clinic Foundation, Cleveland, Ohio, United States